CLINICAL TRIAL: NCT02526108
Title: Energy Expenditure of High Intensity Functional Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002608
Record Dates: First submitted 2015-08-12; First posted 2015-08-18 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIFT (Experimental): High Intensity Functional Training group exercise session. Each session is 45 minutes. Participants will be asked to complete 3 sessions.
  Interventions: Other: HIFT

INTERVENTIONS:
Other: HIFT — Workout alternates short periods of intense exercise using varied, multiple-joint movements, with less-intense active recovery periods. Workout sessions will be led by a trained instructor.
  Other Names: High Intensity Functional Training

SUMMARY:
The purpose of this study is to assess the energy expenditure and intensity of a High Intensity Functional Training (HIFT) session in overweight and obese adult men and women.

DETAILED DESCRIPTION:
High Intensity Functional Training (HIFT), which alternates short periods of intense exercise using varied, multiple-joint movements, with less-intense active recovery periods, may offer an attractive, time efficient alternative to traditional aerobic exercise. Variations of HIFT such as Cross Fit, home workout videos (ie.P90x and Insanity), and boot-camp style group exercise classes have become increasingly popular.

The cardiovascular benefits of HIFT have been demonstrated; however, by doing this study researchers hope to get more information regarding the potential effectiveness of HIFT for weight management, such as the actual level of energy expenditure and exercise intensity elicited by a HIFT session.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 25.0 and 39.9
* Currently participating in HIFT (boot-camp) classes at Kirmayer Fitness Center

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Energy expenditure measured using indirect calorimetry | Energy expenditure will be obtained across a 2 week period after each of 3 exercise sessions
  Energy expenditure will be measured using indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Donnelly, Ed.D., Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Willis EA, Szabo-Reed AN, Ptomey LT, Honas JJ, Steger FL, Washburn RA, Donnelly JE. Energy Expenditure and Intensity of Group-Based High-Intensity Functional Training: A Brief Report. J Phys Act Health. 2019 Jun 1;16(6):470-476. doi: 10.1123/jpah.2017-0585. Epub 2019 May 19. PMID 31104545